CLINICAL TRIAL: NCT00002734
Title: PHASE I STUDY OF INTERFERON ENHANCED INTRAPERITONEAL RADIOIMMUNO-CHEMOTHERAPY FOR OVARIAN CANCER
Brief Title: Radiolabeled Monoclonal Antibody, Paclitaxel, and Interferon Alfa in Treating Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02240; UAB-9502; NCI-B95-0003; CDR0000064633 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2001-02

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Interferon-alpha; Drug Therapy; Paclitaxel; Topotecan

ARMS (1):
- Arm I (Experimental): Patients receive interferon alfa subcutaneously on days 1, 3, 5, and 7; paclitaxel intraperitoneally (IP) on day 4 or topotecan IP on day 6; and 177Lu-CC49 IP on day 6. Treatment continues every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-5 patients receive escalating doses of paclitaxel and decreasing doses of 177Lu-CC49 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 5 patients experience dose limiting toxicity. Once the MTD of paclitaxel is determined, the dose of 177Lu-CC49 is escalated. Once the MTD of 177Lu-CC49 is determined, 90Y-CC49 is substituted. The MTD of 90Y-CC49 is then determined when administered with paclitaxel. Topotecan is then substituted for paclitaxel (administered with the MTD of 177Lu-CC49 and interferon alfa only) and escalated until the MTD is determined.
  Interventions: Biological: recombinant interferon alfa; Drug: chemotherapy; Drug: paclitaxel; Drug: topotecan hydrochloride; Radiation: lutetium Lu 177 monoclonal antibody CC49; Radiation: yttrium Y 90 monoclonal antibody CC49

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: chemotherapy
Drug: paclitaxel
Drug: topotecan hydrochloride
Radiation: lutetium Lu 177 monoclonal antibody CC49
Radiation: yttrium Y 90 monoclonal antibody CC49

SUMMARY:
Phase I trial to study the effectiveness of radiolabeled monoclonal antibody, paclitaxel, and interferon alfa in treating patients who have ovarian cancer. Radiolabeled monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interferon may interfere with the growth of cancer cells. Combining monoclonal antibody, chemotherapy, and interferon alfa may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of intraperitoneal paclitaxel and topotecan when administered as a radiosensitizer prior to intraperitoneal lutetium Lu 177 monoclonal antibody CC49 (177Lu-CC49) following subcutaneous interferon alfa-2b (IFN-A) in patients with persistent or recurrent ovarian cancer.

II. Determine the toxicity associated with intraperitoneal paclitaxel and topotecan in these patients.

III. Examine the conjugate stability, pharmacokinetics, and biodistribution of 177Lu-CC49 given 48 hours after intraperitoneal paclitaxel.

IV. Determine the effects of IFN-A and intraperitoneal paclitaxel on 177Lu-CC49 tumor localization and dosimetry estimates compared to a prior trial with 177Lu-CC49 alone.

V. Determine the MTD of yttrium Y 90 monoclonal antibody CC49 (90Y-CC49) when administered with IFN-A and the dose of paclitaxel used at the MTD level of IFN-A, paclitaxel, and 177Lu-CC49.

VI. Monitor any antitumor effects of this treatment in these patients.

OUTLINE: This is a dose escalation study of paclitaxel, topotecan, lutetium LU 177 monoclonal antibody CC-49 (177Lu-CC49), and yttrium Y 90 monoclonal antibody CC49 (90Y-CC49).

Patients receive interferon alfa subcutaneously on days 1, 3, 5, and 7; paclitaxel intraperitoneally (IP) on day 4 or topotecan IP on day 6; and 177Lu-CC49 IP on day 6. Treatment continues every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-5 patients receive escalating doses of paclitaxel and decreasing doses of 177Lu-CC49 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 5 patients experience dose limiting toxicity. Once the MTD of paclitaxel is determined, the dose of 177Lu-CC49 is escalated. Once the MTD of 177Lu-CC49 is determined, 90Y-CC49 is substituted. The MTD of 90Y-CC49 is then determined when administered with paclitaxel. Topotecan is then substituted for paclitaxel (administered with the MTD of 177Lu-CC49 and interferon alfa only) and escalated until the MTD is determined. Patients are followed at 6 weeks and then every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the ovary or papillary serous carcinoma of extraovarian origin
* Recurrent or persistent following standard surgery and 1 or 2 chemotherapy regimens (with or without paclitaxel), i.e.: persistent disease or progression after chemotherapy with nodules less than the equivalent of 5 x 5 x 5 cm Recurrent carcinoma (after primary or secondary chemotherapy) detected clinically either by exam or rising CA 125 and with radiographic evidence of disease no greater than the equivalent of 5 x 5 x 5 cm nodules
* Residual disease less than 5 x 5 x 5 cm following reassessment laparotomy
* Microscopic residual disease on reassessment laparotomy after chemotherapy
* Tumor TAG-72 positive by immunoperoxidase staining of original or current tumor blocks
* At least 85% free flow of fluid in peritoneal cavity demonstrated by technetium-99m scan or other imaging within 2 weeks prior to treatment
* No evidence of disease outside the peritoneal cavity other than retroperitoneal lymphadenopathy
* No massive ascites

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-2
* WBC at least 3,500/mm3
* Platelet count at least 125,000/mm3
* Hemoglobin greater than 9 g/dL
* No nucleated RBC or significant teardrop RBC morphology
* Bilirubin less than 1.5 mg/dL
* AST/ALT less than 4 times normal
* Creatinine less than 2.0 mg/dL
* HIV negative
* Hepatitis B surface antigen negative
* No hypersensitivity to paclitaxel, polyoxethylated castor oil, or topotecan
* No other malignancy in past 5 years except basal cell skin carcinoma
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior biologic therapy and recovered
* No prior monoclonal antibody therapy
* No concurrent immunotherapy
* No prior bone marrow or stem cell transplantation
* At least 3 weeks since prior chemotherapy (6 weeks since nitrosoureas or mitomycin) and recovered
* No concurrent chemotherapy
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to the abdominal cavity
* No concurrent radiotherapy
* At least 3 weeks since prior major surgery and recovered
* No prior intraperitoneal therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1996-03; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruby F. Meredith, MD, PhD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States

REFERENCES:
- [Result] Meredith R, Alvarez R, Khazaeli MB, et al.: Intraperitoneal radioimmunotherapy for refractory epithelial ovarian cancer with Lu-CC49. Minerva Biotechnologica 10: 100-107, 1998.